CLINICAL TRIAL: NCT05652101
Title: Study of Adaptative Skills and Neurodevelopmental Trajectory for Patients With Hyperekplexia (Startle Disease)
Brief Title: Hyperekplexia : Adaptative Skills and Neurodevelopmental Trajectory
Acronym: StarDev
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0568; 2022-A02107-36 (Other: ID-RCB)
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Hyperekplexia
Keywords: Hyperekplexia; Neurodevelopment trajectory; Adaptative skills
MeSH Terms: conditions — Hyperekplexia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients suffering from hereditary hyperekplexia, above 2 years of age: 40 patients suffering from hereditary hyperekplexia will be included. The investigators study patients suffering from hereditary hyperekplexia. The diagnostic is clinical, based on the following symptoms, appearing shortly after birth: stiffness, exaggerating response startles to unexpected stimuli, generalized stiffness after the startles.
  Children above 2 years old and adults are included, so the neurodevelopment can be evaluated.
  Interventions: Other: collection of medical data; Other: Vineland Adaptive Behaviour Scales (VABS2) questionnaire

INTERVENTIONS:
Other: collection of medical data — The data collected concerns:
  * Sex
  * Age
  * Socio-professional category of patients or parents / level of education of the parents
  * Family history
  * Neonatal patient data (pregnancy, childbirth)
  * Clinical data (age of onset of symptoms, evolution of these symptoms over the years, psychomotor development, schooling, learning difficulties, rehabilitation)
  * Therapeutic data (treatments tried, their dosage and effectiveness, changes in dosage over the years)
  * Paraclinical examinations (Magnetic Resonance Imaging (MRI), scanner, Electroencephalography (EEG))
  * Genetic data if available
Other: Vineland Adaptive Behaviour Scales (VABS2) questionnaire — This is a standardized semi structured interview that measures adaptative skills in 4 areas, in the fields of communication, socialization, daily living, and motricity (for children under 7 years). It can be used for children and adults.
  Rating: 2 = yes, usually, 1 = sometimes or partly, 0 = no, never, N = not applicable (when a child is not yet of sufficient age, for example), NS = don't know. The results by domain and by sub-domain are given in raw scores which are then transformed into equivalent ages using a grid provided for this purpose.

SUMMARY:
Hereditary hyperekplexia is a rare neuronal disorder, caused by genetic defects leading to dysfunction of glycinergic neurotransmission.

The clinical presentation is characterized by stiffness and exaggerated startle responses to unexpected stimuli, that appear shortly after birth.

The generalised stiffness can lead to apnea and sudden infant death syndrome.

Several genes are known to be associated with hereditary hyperekplexia. The most frequent are Glycine Receptor Alpha 1 (GLRA1), Glycine Receptor Beta (GLRB) and Solute Carrier Family 6 Member 5 (SLC6A5). They encode for the postsynaptic glycine receptor (GLRA1, GLRB) and the presynaptic glycine transport (SLC6A5). Genetic mutations in these genes lead to dysfunction in the glycinergic inhibitory neurotransmission.

The neurodevelopment was initially described as normal, or as delayed due to the motor difficulties. Global development delay and intellectual disability are reported as well, in the most recent studies.

Nevertheless, the degree of severity of the learning difficulties and the adaptive faculties of the patients is not specified.

Similarly, the efficacy of clonazepam in hyperekplexia is well known, but the evolution of dosage over time and the frequency of complete withdrawal have never been studied.

The primary endpoint of this study is to describe adaptive skills using a standardized questionnaire, Vineland Adaptive Behavior Scale (VABS2).

Secondary endpoints are:

* Neurodevelopmental course study
* Description of the evolution of the clinical manifestations over the years
* Evaluation of the efficacity of the treatment CLONAZEPAM, initially and over time, and evolution of the dosage
* Comparison of clinical and therapeutical characteristics according to the genotype

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnostic criteria for hyperekplexia (see Thomas et al. BRAIN, 2013):

  * The presence of hypertonia (either hypertonia on examination, axial or segmental, or access of stiffness)
  * Exaggerated reflex startles, to auditory, tactile or visual stimuli
  * The presence of reflex bursts on percussion of the midline
* Children >2 years and adults
* No opposition of one of the two parents (or legal representative) or of the adult patient

Exclusion Criteria:

* The presence of a cause secondary to the hyperekplexia (traumatic, autoimmune, etc.)
* The presence of another cause for a delay in psychomotor development (other neurological pathology, serious head trauma, etc.)
* Pregnant or breastfeeding women
* Person deprived of liberty by judicial or administrative decision

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population of patients followed in pediatric neurology or neurology, for hereditary hyperekplexia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
VABS2 total score and specific scores (socialization, communication, daily living and motricity) | maximum 2 months after the inclusion
  The VABS2 measures adaptative scores in the fields of :
  * Communication (receptive, expressive, written)
  * Daily Living Skills (personal, domestic and in community)
  * Socialisation (interpersonal relationships, play and leisure time, coping skills)
  * Motor Skills (gross and fine motor) for children under 7 years.
  The domains are made up of subdomains in which the scores are added to form the domain composite scores. The four domain composite scores then combine to form the adaptive behaviour composite for those individuals aged birth to 6 years 11 months. Three domain composite scores (communication, daily living skills and socialization) combine to form the adaptive behaviour composite for those aged 7 through 90.
  The results are expressed with standard scores, percentile ranks, adaptive levels and age equivalents.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Femme Mère Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: No